CLINICAL TRIAL: NCT07108933
Title: Effect of Scheduled Autologous Platelet-rich Plasma Guided Injection in the Healing Process of Critical-sized Maxillary Bony Defects After Surgical Excision of Non- Malignant Lesions: A Prospective Randomized Clinical Trial.
Brief Title: Scheduled Autologous PRP Guided Injection in the Maxillary Bony Defects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Horus University (Other)
Responsible Party: Principal Investigator, Eman Abdel Salam Yousef, Associate professor, Horus University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRP in maxillary bone defects
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Bony Defect
Keywords: Platelet-rich plasma, scheduled injection, healing process

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial (RCT)
Masking Description: No masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Injection (Other): Scheduled injection of autologous platelet-rich plasma
  Interventions: Biological: Autologous platelet-rich plasma

INTERVENTIONS:
Biological: Autologous platelet-rich plasma — Guided injection of PRP in bony cavities of maxilla after surgical excision of non-malignant tumors.
  Other Names: PRP

SUMMARY:
Scheduled autologous platelet-rich plasma guided injection is done in critical-sized maxillary bony defects after surgical excision of non- malignant lesions.

DETAILED DESCRIPTION:
The study aims to detect the effect of scheduled autologous platelet-rich plasma- guided injection in the healing process of critical-sized maxillary bony defects after surgical removal of non-malignant lesions by using bone volumetric analysis and density measuring with cone beam computed tomography.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years (adults within a specific age range).

Diagnosis: Non-malignant maxillary bony defects (e.g., benign tumors or cysts).

Health: Generally healthy participants who can tolerate surgery.

Platelet Function: No platelet disorders or blood-related conditions.

Willingness: Informed consent and ability to follow the protocol.

No Use of Blood Thinners: No current use of anticoagulants like aspirin.

Exclusion Criteria:

* Age: Children (under 18) and elderly (over 75).

Malignant Lesions: Participants with cancer or pre-cancerous conditions.

Systemic Illness: Severe conditions (e.g., uncontrolled diabetes, autoimmune disorders).

Platelet Disorders: Low platelet count or bleeding disorders (e.g., hemophilia).

Infections: Active infections or inflammatory conditions (e.g., periodontal disease).

Pregnancy: Women who are pregnant or breastfeeding.

Recent Surgery/Trauma: Recent maxillary surgery or trauma.

Uncontrolled Medications: Use of blood thinners, NSAIDs, or immunosuppressive drugs.

Non-compliance: Unwillingness or inability to follow-up with the protocol.

Substance Abuse: Active drug or alcohol abuse.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Volume of the injected bony defect | after 3 months
  the volume of the injected bony defect is measured by Cone beam computed tomography in millimeters cubic.

SECONDARY OUTCOMES:
Bone density at the injected site | after 3 months
  the density of bone formed at the injected site is measured by Cone beam computed tomography in Hounsfield unit.

CONTACTS AND LOCATIONS:
Overall Officials: Eman Abdel Salam, Prof, Study Director — Head of department of Oral Surgery
Locations (1):
- Dental clinics of Aswan University Hospital, Aswān, Egypt